CLINICAL TRIAL: NCT04942977
Title: Prevention and Rehabilitation After Acute Coronary Syndrome: a New Telemonitoring Strategy
Brief Title: Rehabilitation After Acute Coronary Syndrome: a New Telemonitoring Strategy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catcronic Salut SL (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TSB2014; 484/14/EC (Other: Other)
Record Dates: First submitted 2021-06-12; First posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Angina, Unstable; Non-ST-Segment Elevation Myocardial Infarction (NSTEMI); ST-segment Elevation Myocardial Infarction (STEMI)
Keywords: mobile health; monitoring; cardiac rehabilitation; telerehabilitation; secondary prevention
MeSH Terms: conditions — Angina, Unstable; Non-ST Elevated Myocardial Infarction; ST Elevation Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: Phase III clinical trial, feasibility, controlled and randomized, with two arms: cardiac telerehabilitation (intervention group) and centre-based cardiac rehabilitation (control group)
Who Masked: Care Provider
Masking Description: The characteristics of the interventions do not allow the study to be blinded either for the patient or for the professional. However, the analyses, stress tests and shuttle tests will be performed in a masked manner without the assigned group being identified by the investigators who carry out the examinations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cardiac tele-rehabilitation (Experimental): Patients in the Intervention Group will come to the hospital 4 times during two consecutive weeks, undergoing physical exercise sessions and the same educational talks as in the control group. Subsequently, they will follow the scheduled physical activities and adherence to the risk factor management according to individualised guidelines in their App, until the end of the study period. All data generated are recorded on the professional website. The degree of compliance with the objectives set is monitored by means of 7 coloured icons, which vary according to the target achievement.
  Interventions: Device: telemonitoring
- Centre-based cardiac rehabilitation (Active Comparator): Patients in the control group will come to the hospital 16 times during eight weeks for cycling and muscle strengthening exercises. Educational talks will be given. At the end of the hospital phase, a conventional outpatient follow-up by primary care and the corresponding specialist will be carried out.
  Interventions: Other: Centre-based cardiac rehabilitation

INTERVENTIONS:
Device: telemonitoring — The system consists of the following elements:
  1. Professional website at the hospital, which allows:
     * To set up an individualised care plan
     * To establish the patient's risk profile and targets for improvement.
     * Long-term monitoring of the evolution of cardiovascular risk factors and events that occurred
     * Advise the patient on self-management strategies.
  2. Mobile application software with the following functions:
     * Scheduled exercise sessions
     * Medication reminder
     * Measurement reminder (weight, blood pressure, heart rate, waist circumference, etc.)
     * Messages: Inbox folder for system messages and messages generated by professionals for a specific patient or video conference.
     * Training monitor: guides the patient in the performance of their exercise.
     * Access to certified health information for patients
  Arms: Cardiac tele-rehabilitation
Other: Centre-based cardiac rehabilitation — The physical activity consisted of a workout routine and aerobic cycling training. Patients are instructed to perform 150 minutes per week of moderate physical activity when the hospital phase finishes.
  Arms: Centre-based cardiac rehabilitation

SUMMARY:
Cardiac rehabilitation after an acute coronary syndrome is recognised in the latest guidelines and recommendations published by the major scientific societies as a class I indication. Despite this evidence, the number of patients entering such programmes in Europe is still around 30%. The present study aims to validate a new comprehensive Telerehabilitation System to provide support for cardiac rehabilitation, to optimize it and to test its usefulness in terms of improving adherence to physical exercise and cardiovascular risk parameters.

DETAILED DESCRIPTION:
To validate this approach, a clinical trial was designed to compare a 10-month program of cardiac telerehabilitation with a conventional 8-week centre-based cardiac rehabilitation. Seventy patients will be randomized 1:1 to cardiac telemonitoring or centre-based cardiac rehabilitation. The characteristics of the interventions do not allow the study to be blinded to the patient or the professional. However, the analyses, stress tests and questionaires will be carried out in a masked form without the assigned group being identified by the researchers carrying out the examinations. Assessment for primary and main secondary outcomes will be performed at baseline and at ten months of follow-up, and will include self-reported physical activity (IPAQ), VO2max, blood test, general emotional distress, Adherence to the Mediterranean Diet, quality of life, vital signs, returning to work. The hypothesis is that patients randomised to prolonged telemonitoring will demonstrate higher levels of physical activity at 10-month follow-up, compared to patients in the centre-based cardiac rehabilitation programme, as well other positive changes in the cardiovascular risk profile.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Patients after uncomplicated acute coronary syndrome of both sexes.
* Patients completing a maximal or symptom-limited CPET without angina or electrical ischaemia.
* Age equal to or less than 72 years.

Exclusion Criteria:

* Refusal of informed consent
* Advanced biological age.
* Kidney failure (GFR < 30ml/min/1.73 m2).
* Liver failure (GOT >2 times normal value).
* Ejection fraction less than 50%.
* Uncontrolled blood pressure (>140/90 mmHg).
* Uncontrolled heart failure.
* Dissecting aortic aneurysm.
* Uncontrolled ventricular tachycardia or other dangerous ventricular arrhythmias.
* Aortic or mitral valve disease.
* Recent systemic or pulmonary embolism.
* Active or recent thrombophlebitis.
* Acute infectious diseases.
* Uncontrolled supraventricular arrhythmias or tachycardia.
* Repeated or frequent ventricular ectopic activity.
* Moderate pulmonary hypertension.
* Ventricular aneurysm.
* Uncontrolled diabetes, thyrotoxicosis, myxedema,
* Conduction disorders such as: complete atrioventricular block. Left bundle branch block.
* Wolf-Parkinson-White syndrome.
* Fixed rate pacing.
* Severe anaemia.
* Psychoneurotic disorders.
* Neuromuscular, musculoskeletal and arthritic disorders that may limit activity. may limit activity.

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2020-12-07 (Actual); Study Completion 2020-12-07 (Actual)

PRIMARY OUTCOMES:
Physical activity derived from the International Physical Activity questionnaire (IPAQ) | 10 months
  self-reported physical activity measured in metabolic equivalents (MET-min/week) Minimum value: 0, maximum value 19,278. Higher scores mean a better outcome.

SECONDARY OUTCOMES:
Maximal oxygen uptake | 10 months
  Maximal oxygen uptake during the final 30 seconds of the cardiopulmonary exercise testing (CPET) (ml/kg/min )
Maximal heart rate | 10 months
  Maximal heart rate at the end of the exercise testing (bpm)
Exercise time | 10 months
  stress test duration (minutes)
Lipid parameters | 10 months
  Total cholesterol (mg/dL), HDL cholesterol (mg/dL), LDL cholesterol (mg/dL), Non-HDL cholesterol (mg/dL), Triglycerides (mg/dL), Apolipoprotein B/Apolipoprotein A-I ratio
Glycosylated haemoglobin | 10 months
  Percentage
Weight | 4 and 10 months
  Kg
Waist circumference | 4 and 10 months
  waist circumference change (cm)
Visceral fat | 4 and 10 months
  Percentage
energy expenditure obtained from the International Physical Activity questionnaire (IPAQ) questionaire | 10 months
  Kcal/week
High level of effort obtained from the International Physical Activity questionnaire (IPAQ) questionaire | 10 months
  Percentage
Total score of Adherence to Mediterranean Diet obtained from the Prevention with Mediterranean Diet questionnaire (PREDIMED). | 10 months
  Units. Minimum value: 0, maximum value: 14. Higher scores mean a better outcome.
High level of Adherence to Mediterranean Diet obtained from the Prevention with Mediterranean Diet questionnaire (PREDIMED) | 10 months
  percentage. Minimum value: 0%, maximum value: 100%. Higher scores mean a better outcome.
Global score of emotional distress obtained from the Hospital Anxiety and Depression Scale (HADS) | 10 months
  Units. Minimum value: 0, maximum value: 14. Lower scores mean a better outcome.
Anxiety subscale of emotional distress obtained from the Hospital Anxiety and Depression Scale (HADS) | 10 months
  Units. Minimum value: 0, maximum value: 7. Lower scores mean a better outcome.
Depression subscale of Emotional distress obtained from the Hospital Anxiety and Depression Scale (HADS) | 10 months
  Units. Minimum value: 0, maximum value: 7. Lower scores mean a better outcome.
Global index of the health-related quality of life obtained from the European Quality of Life questionnaire (EuroQol-5D) | 10 months
  Units. Minimum value: 0, maximum value: 1. Higher scores mean a better outcome.
Health status obtained from the European Quality of Life questionnaire (EuroQol-5D) | 10 months
  Units. Minimum value: 0, maximum value: 100. Higher scores mean a better outcome.
smoking cessation | 10 months
  percentage
Time to start the rehabilitation programme after discharge from hospital | 10 months
  days
Returning to work | 10 months
  days
Pulse wave velocity | 10 months
  m/s
User's experience from the System Usability Scale (SUS) score | 10 months
  Units. Minimum value: 0, maximum value: 100. Higher scores mean a better outcome.
Cost-effectiveness analysis | 10 months
  net cost divided by changes in health outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Ernesto Dalli Peydró, MD, Principal Investigator — Hospital Arnau de Vilanova. Valencia
Locations (2):
- Spain (2):
  - Ernesto Dalli Peydró, Valencia
  - Hospital Politécnico Universitario La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ambrosetti M, Abreu A, Corra U, Davos CH, Hansen D, Frederix I, Iliou MC, Pedretti RFE, Schmid JP, Vigorito C, Voller H, Wilhelm M, Piepoli MF, Bjarnason-Wehrens B, Berger T, Cohen-Solal A, Cornelissen V, Dendale P, Doehner W, Gaita D, Gevaert AB, Kemps H, Kraenkel N, Laukkanen J, Mendes M, Niebauer J, Simonenko M, Zwisler AO. Secondary prevention through comprehensive cardiovascular rehabilitation: From knowledge to implementation. 2020 update. A position paper from the Secondary Prevention and Rehabilitation Section of the European Association of Preventive Cardiology. Eur J Prev Cardiol. 2021 May 14;28(5):460-495. doi: 10.1177/2047487320913379. PMID 33611446
- [Background] Thomas RJ, Beatty AL, Beckie TM, Brewer LC, Brown TM, Forman DE, Franklin BA, Keteyian SJ, Kitzman DW, Regensteiner JG, Sanderson BK, Whooley MA. Home-Based Cardiac Rehabilitation: A Scientific Statement From the American Association of Cardiovascular and Pulmonary Rehabilitation, the American Heart Association, and the American College of Cardiology. Circulation. 2019 Jul 2;140(1):e69-e89. doi: 10.1161/CIR.0000000000000663. Epub 2019 May 13. PMID 31082266
- [Background] Frederix I, Vanhees L, Dendale P, Goetschalckx K. A review of telerehabilitation for cardiac patients. J Telemed Telecare. 2015 Jan;21(1):45-53. doi: 10.1177/1357633X14562732. Epub 2014 Dec 4. PMID 25475219
- [Background] Scherrenberg M, Falter M, Dendale P. Providing comprehensive cardiac rehabilitation during and after the COVID-19 pandemic. Eur J Prev Cardiol. 2021 May 14;28(5):520-521. doi: 10.1093/eurjpc/zwaa107. No abstract available. PMID 33623986
- [Background] Reibis R, Salzwedel A, Abreu A, Corra U, Davos C, Doehner W, Doherty P, Frederix I, Hansen D, Christine Iliou M, Vigorito C, Voller H; Secondary Prevention and Rehabilitation of the European Association of Preventive Cardiology (EAPC). The importance of return to work: How to achieve optimal reintegration in ACS patients. Eur J Prev Cardiol. 2019 Sep;26(13):1358-1369. doi: 10.1177/2047487319839263. Epub 2019 Apr 10. PMID 30971111
- [Background] Frederix I, Hansen D, Coninx K, Vandervoort P, Vandijck D, Hens N, Van Craenenbroeck E, Van Driessche N, Dendale P. Medium-Term Effectiveness of a Comprehensive Internet-Based and Patient-Specific Telerehabilitation Program With Text Messaging Support for Cardiac Patients: Randomized Controlled Trial. J Med Internet Res. 2015 Jul 23;17(7):e185. doi: 10.2196/jmir.4799. PMID 26206311